CLINICAL TRIAL: NCT02638181
Title: The Expression of Matrix Metalloproteinase 13（MMP13）, Tissue Inhibitor of Metalloproteinases 3（TIMP13）, and Calcium-sensing Receptor（CaSR） in Human Trabecular Meshwork
Brief Title: The Expression of Matrix Metalloproteinase 13, Tissue Inhibitor of Metalloproteinases 3, and Calcium-sensing Receptor in Human Trabecular Meshwork
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lv Yingjuan (Other)
Responsible Party: Sponsor-Investigator, Lv Yingjuan, department of ophthamology, Tianjin Medical University Eye Hospital
Organization: Tianjin Medical University Eye Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: tjykdxykyy3
Record Dates: First submitted 2015-12-14; First posted 2015-12-23 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Open-angle Glaucoma
Keywords: matrix metalloproteinase 13; tissue inhibitor of metalloproteinases 3; calcium-sensing receptor; trabecular meshwork; open-angle glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- trabeculectomy (Experimental)
  Interventions: Procedure: trabeculectomy

INTERVENTIONS:
Procedure: trabeculectomy

SUMMARY:
This study was to assess the distinct expression of matrix metalloproteinase 13,tissue inhibitor of metalloproteinases 3, and calcium-sensing receptor, in human trabecular meshwork between normal and glaucomatous eyes.The expressions of matrix metalloproteinase 13, tissue inhibitor of metalloproteinases 3 and calcium-sensing receptor in the trabecular meshwork tissues were examined by streptavidin-peroxidase immunohistochemical staining method and western blot, and histological changes of trabecular meshwork were studied by Hematoxylin and Eosin staining.

ELIGIBILITY:
Inclusion Criteria:

* intraocular pressure greater than 22 mmHg with two or more medications
* wide anterior chamber angle
* glaucomatous optic neuropathy (Glaucomatous optic nerve damage was defined as cup-to-disc ratio higher than 0.7 or focal loss of the nerve fiber layer (notch) associated with a consistent glaucomatous visual field defect
* visual field loss consistent with optic nerve damage and visual fields were performed by using standard automated perimetry

Exclusion Criteria:

* the presence of any secondary form of glaucoma including exfoliation syndrome or a history of ocular trauma, etc

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
the expressions of matrix metalloproteinase 13 and calcium-sensing receptor | one hour after operation

SECONDARY OUTCOMES:
histological changes of trabecular meshwork | one hour after operation

CONTACTS AND LOCATIONS:
Overall Officials: xiaorong li, Study Director — Tianjin Medical University Eye Hospital
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China